CLINICAL TRIAL: NCT04815915
Title: Effects of Graston Technique in Patients With Non Specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Principal Investigator, Maryam Shabbir, Associate Professor, Riphah International University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PT-MARYAM SHABBIR-1061
Record Dates: First submitted 2021-03-24; First posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Back Pain
Keywords: Low Back Pain,Pain Numeric Rating Scale,Owestry Disability Index
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental): Graston tool was used to treat patients 3 times in a week according protocol for 6 weeks' treatment plan with extensions bised exercises protocol following pattern of APTA.
  Interventions: Other: Graston technique

INTERVENTIONS:
Other: Graston technique — Graston tool was used to treat patients 3 times in a week according protocol for 6 weeks' treatment plan with extensions bised exercises protocol following pattern of APTA.

SUMMARY:
Non-specific low back pain upsets individuals of all age gathering and is a most significant provider to illness load everywhere on the world. Overseeing rules prescribe emergency to locate the uncommon instances of low back pain that are brought about by actually genuine pathology, thus need demonstrative work-up or proficient arrangement, or both. Since non-specific low back pain doesn't have a known pathoanatomical cause and treatment accentuations on diminishing in agony and its meanings.

To determine the impacts of Graston technique in patients with non-specific low back pain.

This examination was Quasi Experimental study and on the basis of inclusion standards, 20 patients were involved. PNRS and ODI used to collect the data. Graston tool was used to treat patients 3 times in a week according protocol for 6 weeks' treatment plan with extensions bised exercises protocol following pattern of APTA. The data was analyzed using SPSS 21.

ELIGIBILITY:
Inclusion Criteria:

* • Both genders

  * Age (20-40 years)
  * Patients with non-specific backache
  * Trigger points and tender points at low back region

Exclusion Criteria:

* • Patients with chronic diseases

  * Degenerative changes in spine
  * Open wounds around the area to be treated
  * High blood pressure
  * Diabetic neuropathy
  * Cancer (depending on the type and location)
  * Taking anti-coagulants
  * Pregnancy

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-04-05 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
PNRS | 2 months
  Pain Numeric Rating Scale (PNRS) scores in subjects with moderate/severe pain at baseline. *P < 0.0001 vs. baseline. Includes only subjects with baseline PNRS score of 4 to 10. Scale ranges from 0 to 10. Data are shown as mean ± 95% confidence interval. n = 329 for all visits, all with a baseline PNRS score of 4 to 10.
OSWESTRY DISABILITY INDEX | 2 months
  Each section is scored on a 0-5 scale, 5 representing the greatest disability. The index is calculated by dividing the summed score by the total possible score, which is then multiplied by 100 and expressed as a percentage. Thus, for every question not answered, the denominator is reduced by 5

CONTACTS AND LOCATIONS:
Overall Officials: Iqra ZakaUllah, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maher C, Underwood M, Buchbinder R. Non-specific low back pain. Lancet. 2017 Feb 18;389(10070):736-747. doi: 10.1016/S0140-6736(16)30970-9. Epub 2016 Oct 11. PMID 27745712
- [Background] Koch C, Hansel F. Non-specific Low Back Pain and Postural Control During Quiet Standing-A Systematic Review. Front Psychol. 2019 Mar 22;10:586. doi: 10.3389/fpsyg.2019.00586. eCollection 2019. PMID 30967811
- [Background] Balague F, Mannion AF, Pellise F, Cedraschi C. Non-specific low back pain. Lancet. 2012 Feb 4;379(9814):482-91. doi: 10.1016/S0140-6736(11)60610-7. Epub 2011 Oct 6. PMID 21982256
- [Background] Chenot JF, Greitemann B, Kladny B, Petzke F, Pfingsten M, Schorr SG. Non-Specific Low Back Pain. Dtsch Arztebl Int. 2017 Dec 25;114(51-52):883-890. doi: 10.3238/arztebl.2017.0883. PMID 29321099
- [Background] Lakke SE, Soer R, Takken T, Reneman MF. Risk and prognostic factors for non-specific musculoskeletal pain: a synthesis of evidence from systematic reviews classified into ICF dimensions. Pain. 2009 Dec 15;147(1-3):153-64. doi: 10.1016/j.pain.2009.08.032. Epub 2009 Oct 2. PMID 19800735
- [Background] Hayden JA, van Tulder MW, Malmivaara A, Koes BW. Exercise therapy for treatment of non-specific low back pain. Cochrane Database Syst Rev. 2005 Jul 20;2005(3):CD000335. doi: 10.1002/14651858.CD000335.pub2. PMID 16034851
- [Background] Vanwye WR. Nonspecific low back pain: evaluation and treatment tips. J Fam Pract. 2010 Aug;59(8):445-8. PMID 20714454